CLINICAL TRIAL: NCT06352671
Title: Prospective Long-Term Outcomes of a Standardized Ross Procedure
Acronym: ROSS
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 023-286
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This standardized prospective long-term outcome analysis will help reaffirm these findings via a multicenter patient cohort and describe the best practices/techniques for stabilization of the autograft and right ventricular outflow tract reconstruction.

DETAILED DESCRIPTION:
The optimal approach for aortic valve replacement in adults with an anticipated life expectancy greater than fifteen years remains unclear. Mechanical and bioprosthetic valves, while often used, have specific downfalls. Mechanical valves require lifelong anticoagulation usage and bioprosthetic tissue valves have a limited lifespan. The Ross procedure (pulmonary autograft replacement) is the only operation which replaces the diseased aortic valve with a living substitute. Concerns over increased surgical risk and potential long-term failure have shown decreased use of this procedure. However, recent publications from expert centers have shown, in the current era the Ross procedure can be reliably performed safely and reproducibly in selected patients. This standardized prospective long-term outcome analysis will help reaffirm these findings via a multicenter patient cohort and describe the best practices/techniques for stabilization of the autograft and right ventricular outflow tract reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Ross procedure at Baylor Scott and White The Heart Hospital, Plano, The University of Pennsylvania, The University of Washington, and Northwestern University.

Exclusion Criteria:

* Less than 18 years of age
* Presence of active malignancy
* Pregnant at the time of surgery
* Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients undergoing the Ross procedure at the four institutions of the NARC will be included in this study. The primary study center will be Baylor Scott and White The Heart Hospital. The other member institutions include: The University of Pennsylvania, The University of Washington, and Northwestern University. The investigators estimate to enroll around 20 subjects per year at each institution. This will total 80 subjects per year. The investigators plan to enroll patients for 10 years during the duration of the study. The investigators plan to follow patients for their lifetime.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival of the patient | 1 year, 5 year and 10 year
  The primary endpoint of this study will be survival at 1-, 5-, and 10-year intervals.

SECONDARY OUTCOMES:
Rate of re-hospitalization | 1 year after the procedure
  To identify the safety of the Ross procedure measured in percentage
Rate of peri operative morbidity | 1 year after the procedure
  Will be measured in percentage
Rate of re-operation | 1 year after the procedure
  Will be measured in percentage
Rate of re-intervention | 1 year after the procedure
  will be measured in percentage
NYHA status | 1 year after the procedure
  Will be measured as NYHA class I, II,III, IV
Rate of Patients with Anticoagulant Usage | 1 year after the procedure
  Rate of Patients with Anticoagulant Usage 1 year after procedure.
Rate of Bleeding Events | 1 year after the procedure
  Rate of Bleeding Events
Rate of Post Operative Infection | 1 year after the procedure
  Rate of Post Operative Infection

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Heart Hospital, Plano, Texas, United States

REFERENCES:
- [Background] Catterall F, Ames PR, Isles C. Warfarin in patients with mechanical heart valves. BMJ. 2020 Oct 15;371:m3956. doi: 10.1136/bmj.m3956. No abstract available. PMID 33060144
- [Background] El-Hamamsy I, Toyoda N, Itagaki S, Stelzer P, Varghese R, Williams EE, Erogova N, Adams DH. Propensity-Matched Comparison of the Ross Procedure and Prosthetic Aortic Valve Replacement in Adults. J Am Coll Cardiol. 2022 Mar 1;79(8):805-815. doi: 10.1016/j.jacc.2021.11.057. PMID 35210036
- [Background] Mazine A, David TE, Rao V, Hickey EJ, Christie S, Manlhiot C, Ouzounian M. Long-Term Outcomes of the Ross Procedure Versus Mechanical Aortic Valve Replacement: Propensity-Matched Cohort Study. Circulation. 2016 Aug 23;134(8):576-85. doi: 10.1161/CIRCULATIONAHA.116.022800. Epub 2016 Aug 5. PMID 27496856
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e72-e227. doi: 10.1161/CIR.0000000000000923. Epub 2020 Dec 17. No abstract available. PMID 33332150